CLINICAL TRIAL: NCT03425552
Title: Α Randomized, Two-way, Two-treatment, Two-period, Crossover, Open Label, Laboratory-blind, Comparative Bioavailability Study at Steady State Between Paliperidone 100 mg Prolonged Release Suspension for Injection (Test Product) and Xeplion® 100 mg Prolonged Release Suspension for Injection (Reference Product) Following Multiple Intramuscular Injections (Five Doses in Each Period, One Dose Every 28 Days) Administration to Patients With Schizophrenia Who Are Already Receiving a Stable Regimen of Paliperidone Prolonged Release Suspension Via The Intramuscular Route
Brief Title: A Clinical Study to Evaluate the Bioavailability Between Two Products Containing Paliperidone 100 mg in the Form of a Prolonged Release Suspension for Injection in Patients With Schizophrenia Who Are Already Stabilized in This Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pharmathen S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PAL.100/316
Record Dates: First submitted 2018-01-26; First posted 2018-02-07 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2018-10

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test treatment (Experimental): Paliperidone palmitate extended-release injectable suspension for intramuscular use 156 mg (100 mg of Paliperiodne)
  Interventions: Drug: Paliperidone
- Reference treatment (Active Comparator): Paliperidone palmitate 156 mg (equivalent to Paliperidone 100 mg) extended release injectable suspension
  Interventions: Drug: Paliperidone

INTERVENTIONS:
Drug: Paliperidone — Paliperidone Palmitate extended-release injectable suspension 156 mg (100 mg of Paliperidone)
  Arms: Test treatment
Drug: Paliperidone — Paliperidone Palmitate 156 mg (equivalent to Paliperiodne 100 mg) extended release injectable suspension
  Other Names: Xeplion
  Arms: Reference treatment

SUMMARY:
This clinical study will compare the equivalence of two products containing Paliperidone 100 mg in the form of a prolonged release suspension for injection in patients affected by schizophrenia who are already receiving this treatment. Each patient will receive both products (Test and Reference). In total, each patient will receive 10 doses (five doses of the Test product and five doses of the Reference product; one dose every 28 days). Furthermore, the two products (Test and Reference) will be compared with regard to their safety and tolerability.

DETAILED DESCRIPTION:
This study will be a randomized, two-way, two-treatment, two-period, crossover, open label, laboratory-blind, multiple dose study at steady state, under fasting conditions.

To main purpose of this study is to determine the relative bioavailability of Paliperidone 100 mg prolonged release suspension for injection (Pharmathen S.A, Greece) and Xeplion® (Paliperidone) 100 mg Prolonged Release Suspension for Injection (Janssen Pharmaceutica N.V., Belgium) following multiple Intramuscular Injections (five doses in each period, one dose every 28 days) administration to patients with schizophrenia who are already receiving a stable regimen of paliperidone prolonged release suspension via the intramuscular route.

The secondary objective of this study is to evaluate the safety and tolerability between the two products.

Five injections of Paliperidone 100 mg prolonged release suspension will be administered intramuscularly (in the deltoid muscle) to study patients in each period (one injection every 28 days).

A total of 70 patients will be randomized into two sequences (Test-Reference or Reference-Test).

The doses will be administered to study patients in each period, according to the randomization plan , as clarified in the table below:

Period I Day 0 First dose Day 28 Second dose Day 56 Third dose Day 84 Fourth dose Day 112 Fifth Dose

Period II Day 140 First dose Day 168 Second dose Day 196 Third dose Day 224 Fourth dose Day 252 Fifth Dose

Following up the last dose of each period, a series of blood samples will be collected from each patient in order to determine the bioavailability of the received drug. More specifically, patients will return to the clinical site to give the scheduled PK blood samples on Day 113, Day114, Day 115, Day 116, Day 117, Day 118, Day 119, Day 120, Day 121, Day 122, Day 123, Day 124, Day 125, Day 126, Day 127, Day 128, Day 129, Day 130, Day 132, Day 134, Day 136, Day 138, Day 253, Day 254, Day 255, Day 256, Day 257, Day 258, Day 259, Day 260, Day 261, Day 262, Day 263, Day 264, Day 265, Day 266, Day 267, Day 268, Day 269, Day 270, Day 272, Day 274, Day 276, Day 278 and Day 280.

ELIGIBILITY:
Inclusion Criteria:

* The patient is suffering from Schizophrenia.
* The patient age is > 18 years and < 65 years old (inclusive).
* The patient has a body weight not less than 50 Kg and according to the BMI range (18.5 - 35 Kg/m2), (inclusive)
* The patient has received at least 3 doses of Paliperidone 100 mg Prolonged Release Suspension for Injection within the last 3 months.
* The patient is under fasting conditions (food and drinks) for at least 8 hours on the day of screening.
* The patient is available to volunteer for the entire study duration and is willing to adhere to all protocol requirements.
* The findings of the patient are within the range of clinical acceptability in medical history, physical examination, vital signs, ECG, and laboratory results.
* The legally acceptable representative signed the informed consent form and the patient is able to communicate with the investigator and comprehend study-related procedures.
* The patient agrees to use a condom if he is engaged in sexual activity with a woman of childbearing potential.

A condom is required along with another medically acceptable contraceptive method. Medically acceptable methods of contraception include non-hormonal intrauterine device or double barrier method (condom with foam or vaginal spermicidal suppository, diaphragm with spermicide).

* Female patients may be included but must comply with the following in order to be included:
* Women having the potential to become pregnant can be enrolled only if willing to use a clinically acceptable (i.e. intrauterine device or hormonal contraceptives for at least three months) or a double barrier contraceptive measure (i.e. condom and spermicidal gel or diaphragm and spermicidal gel for at least 14 days) prior to the start of the study and through the study and for 30 days after completion of the study, or
* Surgically sterilized for at least 6 months or
* Menopausal women, for at least 1 year

Exclusion Criteria:

* The patient is pregnant or nursing (lactating) women, where pregnancy is defined as the state of the female after conception and until the termination of gestation, confirmed by a positive urine or serum pregnancy test.
* The patient has any significant or organ abnormality as determined by the principal investigator/sub-investigator.
* The patient has skin abnormalities/irritations at the potential injection site (right or left deltoid) as determined by the Principal Investigator/clinical Sub-Investigator.
* The patient has a medical or surgical condition that might interfere with the absorption, metabolism, or excretion of paliperidone.
* The patient has known allergy to the Paliperidone Palmitate or to any ingredient in the preparation.
* The patient has a history of hypersensitivity to heparin.
* The patient intended to significantly change the smoking habits during the trial (i.e. planned cessation or start of smoking career).
* The patient will consume alcohol or caffeine or related xanthine containing foods or beverages for 48 hours prior to each dosing.
* The patient will consume grapefruit or pomelo-containing beverages and foods within 7 days prior to each dosing.
* The patient has a history of or current compulsive abuse of alcohol (more than 10 drinks weekly) or regular exposure to other substance of abuse.
* The patient is on a special diet (for example the patient is a vegetarian), or dieting (on a weight lowering plan) during the month before the study.
* The patient participated in a comparative bioavailability/ bioequivalence study within the last 90 days before first dose of period I.
* The patient participated in a clinical study within the last 90 days before first dose of period I.
* The patient donated blood or any of its constituents (1 unit or 350 ml) within the last 90 days before first dose of period I.
* The patient has positive testing for HIV I & II and/or Hepatitis B and/or Hepatitis C using ELISA method.
* The patient has positive test for illicit drugs or alcohol before any dose.
* The patient is suffering from severe hepatic impairment.
* The patient is suffering from renal impairment
* Presence or history of clinically significant cardiovascular disease (especially known history of QT prolongation, congenital long QT syndrome, recent acute myocardial infarction, cardiac arrhythmias, or with uncompensated heart failure).
* The patient is receiving medicinal products known to prolong the QT interval, e.g. class 1 Antiarrhythmics (e.g., quinidine, disopyramide, procainamide) and class III antiarrhythmics (e.g. amiodarone, sotalol), antihistamines, antipsychotics known to prolong QT interval, and antimalarials (e.g. mefloquine, quinine), tricyclic antidepressants (eg amitriptyline), tetracyclic antidepressants (eg maprotiline).
* The patient is receiving centrally acting medicinal products e.g. anxiolytics, risperidone, opiates, etc. or alcohol
* The patient is receiving drugs that induce orthostatic hypotension (e,g other antipsychotics, tricyclic).
* The patient is receiving medicinal products known to lower the seizure threshold (e.g. phenothiazines or butyrophenones, tricyclics or SSRIs, tramadol, mefloquine, etc.)
* The patient is receiving carbamazepine (causes decrease in mean steady state Cmax and AUC of Paliperidone)
* The patient has current thoughts of suicide or violent tendencies at screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-03-11 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-05-02 (Actual)

PRIMARY OUTCOMES:
Cmax(ss) | 28 days
  Maximum plasma concentration at steady state
AUC0-τ(ss) | 28 days
  AUC during a dosage interval at steady state
Cτ(ss) | 28 days
  Concentration at the end of the dosing interval at steady state

SECONDARY OUTCOMES:
Cmin(ss) | 28 days
  Minimum plasma concentration at steady state
Fluctuation | 28 days
  (Cmax,ss - Cmin,ss) / Cavg,ss
Tmax(ss) | 28 days
  Time until Cmax(ss) is reached
Number of participants with treatment-related adverse events | 281 days

CONTACTS AND LOCATIONS:
Overall Officials: Lina Sabbah, Study Director — Triumpharma
Locations (3):
- Jordan (3):
  - Al-Esraa Hospital, Amman
  - King Abdullah University Hospital, Ar Ramtha
  - Princes Basma Teaching Hospital, Irbid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Guideline for Good Clinical Practice E6(R2) — http://www.ich.org/fileadmin/Public_Web_Site/ICH_Products/Guidelines/Efficacy/E6/E6_R2__Step_4_2016_1109.pdf